CLINICAL TRIAL: NCT01075477
Title: Naturalistic Prospective Non-interventional Study on Rheumatoid Arthritis (RA) Patients Treated With Rituximab According to Local Treatment Guidelines
Brief Title: An Observational Study on Patients With Rheumatoid Arthritis Treated With MabThera (Rituximab)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22609
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort
  Interventions: Drug: rituximab [Mabthera/Rituxan]

INTERVENTIONS:
Drug: rituximab [Mabthera/Rituxan] — As prescribed by physician

SUMMARY:
This observational study will assess the execution, efficacy and safety of treatment with MabThera in patients with rheumatoid arthritis. Data from patients receiving MabThera according to local treatment guidelines will be collected for 29 months. Target sample size is 100-200 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* rheumatoid arthritis
* treatment with rituximab

Exclusion Criteria:

* unable/unwilling to give informed consent to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis on or commencing treatment with rituximab [MabThera]
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Efficacy: DAS28 | 29 months

SECONDARY OUTCOMES:
Efficacy: TJC, SJC, ESR, HAQ, CRP, patient's assessment (VAS) | 29 months
Safety: serious and non-serious adverse events | 29 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Finland (8):
  - Hämeenlinna
  - Helsinki
  - Joensuu
  - Jyväskylä
  - Paimio
  - Riihimäki
  - Seinäjoki
  - Tampere